CLINICAL TRIAL: NCT01419730
Title: The Effect of High-Dose Vitamin D and Physical Activity on Bone Health in Breast Cancer Patients Receiving Hormonal Therapy
Brief Title: Vitamin D and Physical Activity on Bone Health
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Luke Peppone, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 34834
Record Dates: First submitted 2011-08-11; First posted 2011-08-18 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Bone Metabolism Biomarkers; Bone Mineral Density; Physical Fitness
MeSH Terms: interventions — Cholecalciferol; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vitamin D3 50,000 IU (Active Comparator): Vitamin D3 50,000 IU: Patients will be assigned to receive a daily multivitamin, calcium supplement and 50,000 IU/week of vitamin D for a period of 24 weeks.
  Interventions: Drug: Vitamin D3
- Vitamin D3 50,000 IU and Physical Activity (Active Comparator): Vitamin D3 50,000 IU and Physical Activity: Patients will be assigned to receive a daily multivitamin, calcium supplement, 50,000 IU/week of vitamin D, and a progressive walking and resistance band exercise prescription for a period of 24 weeks.
  Interventions: Drug: Vitamin D3; Behavioral: Physical Activity
- Control (No Intervention): Patients will be assigned to receive a daily multivitamin, calcium supplement, vitamin D placebo, and standard care monitoring.

INTERVENTIONS:
Drug: Vitamin D3 — Vitamin D3 50,000 IU
  Arms: Vitamin D3 50,000 IU; Vitamin D3 50,000 IU and Physical Activity
Behavioral: Physical Activity — Progressive walking and resistance band exercise prescription for a period of 24 weeks
  Arms: Vitamin D3 50,000 IU and Physical Activity

SUMMARY:
This research will examine the effectiveness of vitamin D or placebo (the placebo is a tablet that looks like Vitamin D study drug, but has no Vitamin D study drug in it), with and without physical activity (walking and progressive resistance exercise), in treating bone loss in women who have undergone treatment for breast cancer. The investigators would also like to find out if the physical activity program improves cardiovascular fitness, energy expenditure, muscular strength, muscle mass, and balance. One hundred five (105) subjects are expected to take part in this study. The investigators don't know if bone loss in breast cancer survivors should be treated differently than bone loss in other women.

ELIGIBILITY:
Inclusion Criteria:

* Must be female and have a primary diagnosis of Stage I, II, or III hormone-receptor positive breast cancer.
* Women must be postmenopausal at time of enrollment.
* Must provide informed consent.
* Must be willing to discontinue use of calcium and/or vitamin D supplements.
* Participants must have an ionized serum calcium level within normal limits (1.19-1.29mmol/L) and a total corrected serum calcium of < 10.6 mg/dl.
* Participants must be slightly vitamin D deficient (serum vitamin D level <32ng/ml)
* Must have a functional capacity rating of ≤ 2 on the Eastern Cooperative Oncology Group (ECOG) performance status when assessed at baseline.132
* Must have the approval of their treating physician (or physician's nurse practitioner or physician's assistant) to participate in sub-maximal physiological fitness testing and a low to moderate home-based walking and progressive resistance exercise program and to receive the 24-week supplementation of vitamin D.
* Must be less than five years from the diagnosis of breast cancer and must be within 12 months of starting treatment with aromatase inhibitors (AI) in accordance with American Society of Clinical Oncology (ASCO) guidelines.

Exclusion Criteria:

* Subjects with life-threatening conditions that would preclude them from breast cancer treatment including chronic cardiac failure, which is unstable despite medication use, uncontrolled hypertension, uncontrolled diabetes mellitus, or unstable coronary artery disease.
* Patients who had a myocardial infarction within the past year.
* Patients with severe metabolic disorders, which includes phenylketonuria (PKU), homocystinuria, and Fabry's disease, that would preclude them from taking calcitriol.
* Patients with impaired renal function (CRCL < 60 mL/min) or who had kidney stones (calcium salt) within the past 5 years.
* Patients with hypercalcemia (corrected serum Ca ≥ 10.6 mg/dl) or a history of hypercalcemia or vitamin D toxicity.
* Patients currently taking calcium supplements or aluminum-based antacids must be willing to discontinue their use if they are to enroll in the study.
* Patients currently taking vitamin D supplements must immediately discontinue their use if they are to enroll in the study.
* Patients with a known sensitivity to vitamin D.
* Patients who are severely vitamin D deficient (<10 ng/ml).
* Women on antiresorptive drugs (e.g. bisphosphonates) within the past year.
* Patients not capable of participating in an exercise intervention due to severe knee arthrosis or ligament/cartilage injuries of the lower extremities.
* Women with malabsorptive syndromes (i.e. cystic fibrosis, chronic pancreatitis) or taking medications that decrease the absorption of fat soluble vitamins (i.e. Orlistat, Questran).

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Measure the amount of bone loss in non-metastatic breast cancer patients receiving a high dose vitamin D therapy along with a structured home-based walking and progressive resistance exercise program. | 24 weeks
  To collect preliminary data on the effects of vitamin D therapy and exercise (alone or in combination) on bone metabolism biomarkers in non-metastatic breast cancer patients who began hormonal therapy within the previous 12 months.
  To collect preliminary data on the effects of vitamin D therapy and exercise (alone or in combination) on bone mineral density (BMD) as measured by a dual energy X-ray absorptiometry (DXA) in non-metastatic breast cancer patients who began hormonal therapy within the previous 12 months.

SECONDARY OUTCOMES:
Measure the effect of vitamin D and exercise on physical fitness in non-metastatic breast cancer patients | 24 weeks
  Measuring physical fitness includes balance, aerobic capacity, and muscle strength in non-metastatic breast cancer patients who begin hormonal therapy within the previous 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Luke J Peppone, PhD, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States